CLINICAL TRIAL: NCT02762435
Title: Randomized Controlled Trial of Acupressure to Improve Patient Satisfaction and Quality of Recovery in Hospitalized Patients
Brief Title: Acupressure in Hospitalized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 867005-3
Record Dates: First submitted 2016-04-14; First posted 2016-05-05 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Acupressure
MeSH Terms: interventions — salicylhydroxamic acid; Acupressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- control (Placebo Comparator): No pressure applied to the 3 points
  Interventions: Other: control
- sham (Sham Comparator): Light touch applied to the 3 points (2 minutes each at PC6, LI4, and HT7, three times per day for 2 days)
  Interventions: Other: sham
- acupressure (Experimental): Moderate pressure applied to the 3 points (2 minutes each at PC6, LI4, and HT7, three times per day for 2 days)
  Interventions: Other: acupressure

INTERVENTIONS:
Other: sham — light touch at established points on hand and wrist
  Arms: sham
Other: control — no contact with the subject
  Arms: control
Other: acupressure — moderate pressure at established points on hand and wrist
  Arms: acupressure

SUMMARY:
After written informed consent eligible hospitalized patients will be randomized to one of 3 arms (1:1:1:): control, sham, accupressure (3 points on the hand and wrist three times per day). Quality of recovery and other measures of patient satisfaction will be recorded.

DETAILED DESCRIPTION:
After written informed consent eligible hospitalized patients will be randomized to one of 3 arms (1:1:1:): control (no touch), sham (light touch), acupressure (2 minutes moderate pressure each at PC6, LI4, and HT7 three times per day). Quality of recovery using the validated Quality of Recovery (QOR) 15 score and other measures of patient satisfaction (nausea score, pain score) will be recorded at baseline and after their 6 study sessions.

ELIGIBILITY:
Inclusion Criteria:

1. adults
2. patients at Stony Brook hospital
3. expected to be hospitalized for at least 3 days
4. able to sign informed consent and participate in the study

Exclusion Criteria:

1. Under 18 years of age
2. Do not have access to the 3 points on the hand and wrist due to skin breakdown, ulcers, cellulitis, broken bone, indwelling catheter within 5 cm radius of the pressure points.
3. Significant dementia or altered mental status that would prevent assessment of the QOR survey
4. Allergic reaction to ink
5. Stroke or other neurologic condition which precludes sensation in both upper extremities.
6. Ongoing use of regional anesthetic technique
7. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Recovery score | Time Frame: Day 0, Day 2
  The validated QOR15 score will be assessed at baseline (Day 0) and after the 6 sessions have been completed (Day 2) and the change in QOR15 (Day 2 minus Day 0) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Bennett-Guerrero, MD, Principal Investigator — Stony Brook Medicine
Locations (1):
- Stony Brook Medicine, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Noll E, Shodhan S, Romeiser JL, Madariaga MC, Page C, Santangelo D, Guo X, Pryor AD, Gan TJ, Bennett-Guerrero E. Efficacy of acupressure on quality of recovery after surgery: Randomised controlled trial. Eur J Anaesthesiol. 2019 Aug;36(8):557-565. doi: 10.1097/EJA.0000000000001001. PMID 30985537
- [Derived] Noll E, Shodhan S, Madariaga MC, Page CR, Santangelo D, Guo X, Al Bizri E, Pryor AD, Romeiser J, Bennett-Guerrero E. Randomized trial of acupressure to improve patient satisfaction and quality of recovery in hospitalized patients: study protocol for a randomized controlled trial. Trials. 2017 Mar 7;18(1):110. doi: 10.1186/s13063-017-1839-1. PMID 28270180